CLINICAL TRIAL: NCT06855277
Title: A Phase III, Open-label, Multi-center, Randomized Study Comparing AAA817+ARPI Versus Standard of Care in Adult Participants With PSMA-positive Metastatic Castration Resistant Prostate Cancer
Brief Title: Study Comparing AAA817+ARPI Versus Standard of Care in Adult Participants With PSMA-positive mCRPC
Acronym: AcTFirst
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAA817B12301; 2024-512340-32 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2025-02-18; First posted 2025-03-03 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Prostate Cancer
Keywords: Positive Metastatic Castration Resistant Prostate Cancer; PSMA; PSMA-positive; AAA817; [225AC] AC-PSMA-617; Radioligand Therapy; RLT; Androgen receptor pathway inhibitor; ARPI; Taxane; Metastatic castration resistant prostate cancer; mCRPC; AcTFirst; [177Lu]Lu- PSMA-617; AAA617
MeSH Terms: conditions — Prostatic Neoplasms | interventions — (225)Ac-PSMA-617; enzalutamide; abiraterone; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Investigational Arm: AAA817+ARPI (enzalutamide or abiraterone) (Experimental): Participants will receive AAA817 infusion directly into a vein with ARPIs.
  Interventions: Drug: AAA817; Drug: ARPI
- Investigational Arm: AAA817 (Experimental): Participants will receive AAA817 infusion directly into a vein.
  Interventions: Drug: AAA817
- Control arm: Investigator's choice of SoC (ARPI or chemotherapy or AAA617) (Active Comparator): Participants will receive standard treatment as decided by the trial doctor either as a taxane-based chemotherapy infusion directly into a vein or ARPI change either as capsules or tablets or AAA617 monotherapy infusion directly into a vein.
  Interventions: Drug: ARPI; Drug: Standard of Care

INTERVENTIONS:
Drug: AAA817 — AAA817 is being studied for treating PSMA positive mCRPC. Inside the body, it attaches itself to PSMA on the cell surface of the prostate cancer cells and emits radiation to kill them. This treatment is also called a radioligand therapy.
  Other Names: [225Ac]Ac-PSMA-617
  Arms: Investigational Arm: AAA817; Investigational Arm: AAA817+ARPI (enzalutamide or abiraterone)
Drug: ARPI — Androgen receptor pathway inhibitor (ARPI): An ARPI is approved for the treatment of prostate cancer. It works by blocking signals from male hormones, such as testosterone, that helps cancer cells grow. By blocking these signals, an ARPI slows down or stops the growth of prostate cancer cells. In this trial, participants will be given either enzalutamide or abiraterone.
  Other Names: Enzalutamide or Abiraterone
  Arms: Control arm: Investigator's choice of SoC (ARPI or chemotherapy or AAA617); Investigational Arm: AAA817+ARPI (enzalutamide or abiraterone)
Drug: Standard of Care — Standard treatment includes approved treatment for mCRPC. In this trial, the trial doctor will decide which available treatment participants will receive. The trial doctor will select either an ARPI of enzalutamide or abiraterone, or a taxane based chemotherapy of docetaxel or cabazitaxel or [177Lu]Lu-PSMA-617 (AAA617).
  Other Names: ARPI enzalutamide; ARPI abiraterone; Taxane based chemotherapy of docetaxel; Taxane based chemotherapy of cabazitaxel; [177Lu]Lu-PSMA-617 (AAA617)
  Arms: Control arm: Investigator's choice of SoC (ARPI or chemotherapy or AAA617)

SUMMARY:
The purpose of this study is to determine whether [225Ac]Ac-PSMA-617 (AAA817), given for up to 6 cycles at a dose of 10 Megabecquerel (MBq) +/- 10%, plus androgen receptor pathway inhibitor (ARPI), improves the radiographic progression free survival (rPFS) compared to investigator's choice of standard of care (SOC) (ARPI change or taxane-based chemotherapy or [177Lu]Lu-PSMA-617 (AAA617)) in adult participants with PSMA-positive metastatic castration resistant prostate cancer (mCRPC) treated with another ARPI as last treatment and who have not been exposed to a taxane-containing chemotherapy in the mCRPC setting nor have received any prior PSMA-targeting radioligand therapy.

DETAILED DESCRIPTION:
This is a phase III, open label, multicenter randomized study. The study aims at evaluating the superiority of 225Ac-PSMA-617 combined with androgen receptor pathway inhibitor (ARPI) over a change of ARPI or chemotherapy or [177Lu]Lu-PSMA-617 (AAA617) in prolonging progression free survival (rPFS).

Screening period: At screening, the participants will be assessed for eligibility and will undergo a positron emission tomography (PET)/computed tomography (CT) scan to evaluate PSMA positivity. Only participants with PSMA positive cancer and confirmed eligibility criteria will be randomized.

Participants randomized to the investigational arms will receive up to 6 doses of AAA817 10 Mbq +/- 10% given intravenously with or without an ARPI (oral enzalutamide or oral abiraterone) per investigator's choice. Treatment with ARPI should continue as per protocol end of treatment criteria.

Participants randomized to SoC will be treated with an ARPI change (oral enzalutamide or oral abiraterone) or taxane-based chemotherapy (docetaxel or cabazitaxel) or [177Lu]Lu-PSMA-617 (AAA617)' per investigator's choice. Treatment with ARPI should continue as per protocol end of treatment criteria. Treatment duration with taxane-based chemotherapy or AAA617will depend on the chosen regimen per the investigator's discretion following local guidelines as per standard of care and product labels and adhere to the protocol end of treatment criteria.

Supportive care will be allowed in both arms at the discretion of the investigator and includes available care for the eligible participant according to best institutional practice for mCRPC treatment, including androgen deprivation therapy (ADT).

Safety will be assessed routinely during the study. Crossover is not allowed among study arms.

The study will be conducted in the USA among other countries globally.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Participants must be adults ≥ 18 years of age.
* Participants must have an ECOG performance status of 0 to 2.
* Participants must have histological, and/or cytological confirmation of adenocarcinoma of the prostate. Participants with mixed histology (neuroendocrine) are not eligible.
* Participants who have received taxane-based chemotherapy in mHSPC setting are eligible if they are deemed appropriate for chemotherapy, ARPI change or AAA617 as the next line of therapy in the opinion of the Investigator. Note: Participants who have received taxane-based chemotherapy for mCRPC are excluded.
* Participants must not have received taxane-based chemotherapy in mCRPC setting (allowed in mHSPC setting).
* Participants must have PSMA-PET positive disease using a PSMA imaging agent that is approved as per protocol.
* Participant must have been diagnosed with mCRPC with documented progressive disease while on treatment with ARPI in mHSPC or earlier setting as their last treatment (and did not progress on more than one ARPI).

  * Participants with deleterious or suspected deleterious germline or somatic homologous recombination repair (HRR) gene-mutated metastatic castration-resistant prostate cancer, as per local testing, may be enrolled if they had prior exposure to PARPi.

Key Exclusion Criteria:

* Previous anti-cancer treatment with any approved or investigational radiopharmaceuticals (for example, [177Lu]Lu-PSMA, [177Lu]-DOTA, or Radium- 223.)
* Previous treatment with any external beam radiotherapy including hemi-body radiation within 6 weeks of randomization (within 2 weeks for radiotherapy of localized metastases).

  * Any prior PARP inhibitor or other systemic anticancer therapy administered for metastatic castration-resistant prostate cancer (mCRPC). Any other approved or investigational systemic therapy (including chemotherapy, immunotherapy, biologics, or monoclonal antibodies) is prohibited within 28 days or 5 half-lives (whichever is shorter) before randomization.

Note: Prior ARPI administered in the mHSPC setting or earlier may continue until C1D1.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 940 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-09-29 (Estimated); Study Completion 2032-11-04 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression Free Survival (rPFS) | From the date of randomization to the date of the first documented radiographic disease progression using conventional imaging, or death due to any cause, whichever occurs first, assessed up to approximately 40.0 months.
  Time to radiographic disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) (Key Secondary Endpoint) | From the date of randomization to the date of death due to any cause, assessed up to approximately 40 months.
  Time to death due to any cause.
Radiographic Progression Free Survival by by Prostate Cancer Working Group 3 (PCWG3)-modified RECIST v1.1 (Key Secondary) | From date of randomization to the date of the first documented radiographic disease progression or death due to any cause, whichever occurs first, assessed up to approximately 40.0 months.
  Time to radiographic disease progression, using by blinded independent central review (BICR) using conventional imaging and Prostate Cancer Working Group 3 (PCWG3)-modified RECIST v1.1 criteria or death due to any cause.
Overall Survival in participants with PSMA-positive mCRPC treated with another ARPI. (Key Secondary) | From the date of randomization to the date of death due to any cause.
  Time to death due to any cause.
rPFS in participants treated with AAA817 | From the date of randomization to the date of the first documented radiographic disease progression, or death due to any cause, whichever occurs first, assessed up to approximately 40.0 months.
  rPFS time to the date of first documented radiographic disease progression or death due to any cause, whichever occurs first.
Progression Free Survival (PFS) | From date of randomization to the first documented progression by investigator's assessment or death due to any cause, whichever occurs first, assessed up to approximately 40.0 months.
  Time to first documented progression or death due to any cause.
Progression Free Survival (PFS2) | From date of randomization until date of second progression or date of death from any cause, whichever comes first, assessed up to approximately 40.0 months.
  Time to first documented progression on next line of antineoplastic therapy or death from any cause.
Overall Response Rate (ORR) | From the date of randomization to the date of the first documented radiographic disease progression, or death due to any cause, whichever occurs first, assessed up to approximately 40.0 months.
  The proportion of participants with best overall response (BOR) of confirmed complete response (CR) or partial response (PR) in soft tissue.
Disease Control Rate (DCR) | From the date of randomization to the date of the first documented radiographic disease progression or death due to any cause, whichever occurs first, assessed up to approximately 40.0 months.
  The proportion of participants with BOR of confirmed CR, PR, stable disease (SD) or non-CR/non-progressive disease (PD) in soft tissue.
Duration of Response (DoR) | From the date of first documented response (CR or PR) for confirmed responders and the date of first documented radiographic progression in soft tissue or death due to any cause, whichever occurs first, assessed up to approximately 40.0 months.
  Time between the date of first documented response and the date of first documented radiographic progression or death due to any cause.
Time to first radiographic soft tissue progression (TTSTP) | From the date of randomization to the date of radiographic soft tissue progression or death due to any cause, whichever occurs first, assessed up to approximately 40.0 months.
  Time to radiographic soft tissue progression.
Time to first symptomatic skeletal event (TTSSE) | From the date of randomization to the date of the first documented radiographic disease progression, or death due to any cause, whichever occurs first, assessed up to approximately 40.0 months.
  Time to date of first new symptomatic skeletal event of death due to any cause.
Prostate specific antigen response (PSA50 and PSA90) | From the date of randomization to the date of safety follow up, assessed up to approximately 40.0 months.
  The percentage of participants who achieved ≥ 50% and ≥ 90% decrease from baseline, respectively.
Time-concentration profiles and PK parameters of AAA817 | From Cycle 1 Day 1 up to approximately cycle 5 days 11 (each cycle is 8 weeks).
  Time-concentration profiles and PK parameters of AAA817 (e.g. AUC, Cmax).
Change from baseline on FACT-P Prostate Cancer Subscale (PCS) | From randomization to the first occurrence of worsening on the score or death due to any cause, whichever occurs first, assessed up to approximately 40.0 months.
  Change from baseline on FACT-P Prostate Cancer Subscale (PCS). FACT-P assesses symptoms/problems related to prostate carcinoma and its treatment.
Time to worsening on the Worst Pain | From randomization to the first occurrence of worsening from baseline, or death due to any cause, whichever occurs first, assessed up to approximately 40.0 months.
  Time to worsening on the Worst Pain is defined as the time from randomization to the first occurrence of worsening on the Worst Pain item (BPI-SF) or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (40):
- United States (12):
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Miami Cancer Institute at Bapt, Miami, Florida
  - Univ Of Iowa Hospitals And Clinics, Iowa City, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Wash U School of Medicine, St Louis, Missouri
  - Bassett Medical Center, Cooperstown, New York
  - Weill Cornell Medicine NY-Presb, New York, New York
  - University of Rochester Medical Ctr, Rochester, New York
  - Associated Med Professionals of NY, Syracuse, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology San Antonio, San Antonio, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Adelaide, South Australia
- Novartis Investigative Site, São Paulo, São Paulo, Brazil
- China (9):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Shenyang, Liaoning
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Hong Kong, Hong Kong
- India (2):
  - Novartis Investigative Site, Gurgaon, Haryana
  - Novartis Investigative Site, Mumbai, Maharashtra
- Japan (7):
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Chiba
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kyoto
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Taiwan (2):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com